CLINICAL TRIAL: NCT05322057
Title: Efficacy of Cx601 (Darvadstrocel) for the Treatment of Perianal Fistulizing Crohn's Disease - a Prospective Nationwide Multicentre Study
Brief Title: Efficacy of Cx601 (Darvadstrocel) for the Treatment of Perianal Fistulizing Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Dr. med. univ., Medical University of Vienna
Other Study IDs: 1682/2018
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Crohn Disease; Fistula Perianal
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with Crohn's disease and complex perianal fistula: 14 patients with Crohn's disease refractory to standard treatment for complex perianal fistula got enrolled in this study.
  Interventions: Drug: Darvadstrocel

INTERVENTIONS:
Drug: Darvadstrocel — Injection of 120 million allogeneic expanded adipose-derived mesenchymal stem cells around the fistula opening and around the fistula tract
  Other Names: Alofisel

SUMMARY:
The use of mesenchymal stem cells is considered a novel and promising therapeutic option for patients with perianal fistulizing Crohn's disease. However, due to limited clinical data, this multicentre, nationwide study aimed to assess its clinical efficacy in closing complex anal fistula.

DETAILED DESCRIPTION:
Fifteen applications in 14 patients (3 male, 11 female) with complex anal fistulas treated in three tertiary hospitals in Austria were included between October 2018 and April 2021. Injection of 120 million allogeneic expanded adipose-derived mesenchymal stem cells (Cx601 - Darvadstrocel, Alofisel®) was performed in each patient. Closure of the external fistula opening without secretion by finger compression was defined as success.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 and older who had a non-active or mildly active luminal CD with complex fistula with a maximum of two internal and three external fistulas

Exclusion Criteria:

* rectovaginal fistulas
* rectal and/or anal stenosis
* active proctitis
* diverting stomas
* an abscess (<2cm) that was not drained at the fistula preperation visit

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 14 patients with Crohn's disease and complex fistula got enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Fistula Closure | 1 year
  The study's primary endpoint was established at week 52 with clinically assessed fistula closure.

SECONDARY OUTCOMES:
Evaluation of perianal disease | 1 year
  At every follow up visit the perianal disease was evaluated using the PDAI (Perianal disease activity index)
Evaluation of Crohn's disease | 1 year
  Crohn's disease was evaluated by using the HBI (Harvey Bradshaw Index)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, Prof.MD, Study Chair — Medical University of Vienna, Head of Pelvic Floor Surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD can be shared just in anonymised form in case of an ethical agreement with other researches.